CLINICAL TRIAL: NCT05364788
Title: Characterisation of Appendiceal Cancer by Genomic and Transcriptomic Analysis and Correlation With Clinical Outcomes
Brief Title: Molecular Characterisation of Appendiceal Cancer
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp215
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Appendiceal Cancer
MeSH Terms: conditions — Appendiceal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival Formalin Fixed Paraffin Embedded (FFPE) human tissue from appendix cancer primary tumour and peritoneal metastases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Appendiceal Cancer Patients
  Interventions: Other: Retrospective tissue sample analysis

INTERVENTIONS:
Other: Retrospective tissue sample analysis — Acquisition of archival Formalin Fixed Paraffin Embedded (FFPE) human tissue from appendix cancer primary tumour and peritoneal metastases, which are stored in NHS pathology - taken from standard care biopsies.

SUMMARY:
Patients ≥ 18 years old who have been diagnosed with appendiceal cancer with peritoneal metastases, have had cytoreductive surgery, have availability of archival tumour tissue and have consented to our institutional biobank program or have a waiver of consent for deceased patients who have not had the opportunity to provide biobank consent (requested at the time of ethics review). Descriptive analysis of the proportion of genetic mutations identified in appendiceal cancers. This is given by the percentage of pathogenic mutations in the peritoneal metastasis compared to the primary tumour.

DETAILED DESCRIPTION:
Appendiceal cancer is a rare and understudied cancer that frequently leads to metastatic disease with production of copious gelatinous collections in the abdomen, causing severe illness and poor survival. The only definitive treatment available is a complex and aggressive surgical procedure involving removal of organs and the internal lining of the abdomen. There is an urgent need to define clinical predictors of survival, the role of chemotherapy and to develop new treatments.

The genetics of appendiceal cancer has been reported in small cohorts of patients but there has been limited research on how mutations affect treatments or survival. There is no information on how and why primary appendiceal cancers often spread just to the lining of the abdomen. Understanding how genetic mutations evolve in the tumours are important for working out treatments to prevent the spread of cancer. Current high throughput laboratory techniques for analysing the genetic makeup of appendiceal cancer has the power to identify mutation patterns than might predict for treatments and survival outcomes.

This study proposes completing tumour genetic studies on archived cancer tissue removed routinely from patients who previously have had surgery for their appendiceal tumour. The results of genetic tests can then be compared to clinical characteristics of the patients such as survival time and treatments received. Genes in primary appendix tumours can be compared to those in tumours that have spread into the lining of the abdomen to describe what changes if any occur during the spreading process.

This study will help make progress towards better and personalised treatment options, identifying predictors of treatment success and long-term survival. Improved treatments and better selection of patients may ultimately improve quality of life and help patients live longer.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Patients ≥ 18 years old who have been diagnosed with appendiceal cancer with peritoneal metastases,
2. have had cytoreductive surgery
3. have availability of archival tumour tissue

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with appendiceal cancer with peritoneal metastases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-07-03 (Estimated)

PRIMARY OUTCOMES:
Characterise the genes of appendiceal cancer. | 2 years
  Descriptive analysis of the proportion of genetic mutations identified in appendiceal cancers. This is given by the percentage of pathogenic mutations in the peritoneal metastasis compared to the primary tumour.

SECONDARY OUTCOMES:
Descriptive analysis in proportions | 2 years
  The descriptive difference in proportion of genetic mutations identified in primary appendiceal tumours compared to mutations in peritoneal metastases. Association between molecular subtypes and categorical variables were measured by Fisher's exact or X2 tests. Associations with continuous variables will be evaluated by Kruskal-Wallis tests or ANOVA. Kaplan-Meier methods will calculate survival outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided